CLINICAL TRIAL: NCT01142856
Title: A Single Patient Treatment Protocol for Autologous Mesenchymal Stem Cell Intraspinal Therapy in Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Mesenchymal Stem Cells for Treatment of Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Anthony J. Windebank, M.D., Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-001995
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

INTERVENTIONS:
Biological: autologous mesenchymal stem cells — single intrathecal dose of 10x6 cells by lumbar puncture.

SUMMARY:
The purpose of this study is to determine the safety of injecting mesenchymal stem cells through intraspinal delivery for the treatment of ALS.

DETAILED DESCRIPTION:
A single patient safety study for harvesting, expanding ex vivo and injecting autologous mesenchymal stem cells (MSC's) into the subarachnoid space of a patient with amyotrophic lateral sclerosis (ALS). Cells will be isolated from adipose tissue by subcutaneous biopsy and expanded using an FDA-approved protocol. They will then be injected by lumbar puncture into the cerebrospinal fluid. Injection will be completed in the in- patient clinical research unit (CRU). the patient will be followed for two years.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 years, if female, must be menopausal or had hysterectomy
* resident and citizen of the United States
* history of a chronic onset of a progressive motor weakness
* able to comply with protocol requirements
* can provide written consent

Exclusion Criteria:

* does not have renal disease (Creatine > 2.0)
* does not have active systemic disease
* does not have any clinically significant abnormalities on prestudy laboratory evaluation
* does not have any clinically significant medical condition (e.g.,within 6 months of baseline, had a myocardial infarct, angina pectoris, and/or congestive heart failure), that in the opinion of the investigator, would compromise the safety of the patient
* does not have a history of cancer including melanoma with the exception of localized skin cancers (with no evidence of metastasis, significant invasion,or re-occurrence within 3 years of baseline).
* has not used an investigational drug within 30 days of baseline visit
* does not have a tracheostomy
* does not have a Beck's Depression Inventory score >16

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Safety | 2 year follow-up
  Clinical monitoring of possible reaction to intrathecal MSC delivery including blood pressure, temperature and pain score.

SECONDARY OUTCOMES:
Neurologic disability score | Two year follow-up
  Quantitative, summated, manual muscle testing

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J. Windebank, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States